CLINICAL TRIAL: NCT06475170
Title: Laparoscopic Proximal Gastrectomy With 'λ+α' Double-Tract Reconstruction for Upper-Third Early Gastric Cancer: A Randomized Clinical Trial.
Brief Title: Preliminary Efficacy Analysis of 'λ+α' Double-Tract Reconstruction After Laparoscopic Proximal Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Northern Jiangsu People's Hospital, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NorthernJiangsu1
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Reflux Esophagitis
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- λ+α double-tract anastomosis (Experimental)
  Interventions: Procedure: proximal gastrectomy combined with 'λ+α' double-tract anastomosis
- double-tract anastomosis (Active Comparator)
  Interventions: Procedure: proximal gastrectomy combined with 'λ+α' double-tract anastomosis

INTERVENTIONS:
Procedure: proximal gastrectomy combined with 'λ+α' double-tract anastomosis — 1. The lymphadenectomy is performed according to the Japanese Gastric Cancer Treatment Guidelines
  2. Transection of the esophagus is performed using a linear stapler 2cm away from the proximal end of the tumor.
  3. The jejunum is dissected 30 cm from the flexor ligament and the distal jejunum is lifted in an anterior colonic direction to the esophageal dissection.
  4. Esophagojejunal anastomosis at 16 cm from the distal jejunal stump；
  5. Residual gastrojejunostomy at 8 cm from the distal jejunal stump；

SUMMARY:
The incidence of proximal gastric cancer has increased significantly in recent years. This may be due to weight gain, alcohol consumption, gastroesophageal reflux disease (GERD), and precancerous lesions. With a deeper understanding of the pattern of lymph node metastasis and the emergence of anti-reflux procedures, proximal gastrectomy has gradually received clinical attention. For early-stage upper gastric cancer and esophagogastric combination cancer cases that are expected to have a good prognosis, the ideal surgical procedure should be to preserve the distal stomach to improve the quality of life and to choose a reasonable digestive tract reconstruction method to prevent reflux. The anti-reflux effect of various proximal gastrectomy digestive tract reconstruction methods and the advantages and disadvantages of various surgical procedures are controversial, and the recognized ideal reconstruction method has not yet been established. Therefore, based on the stomach's anatomical features and the intercalated jejunum's anti-reflux mechanism, we propose a true dual-channel anastomosis for GI reconstruction, i.e., the "λ+α dual-channel anastomosis". This study aimed to investigate the efficacy and safety of proximal gastrectomy combined with "λ+α double-channel anastomosis" in the treatment of early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Age between 18-75 years old, male or female; Pathological diagnosis of preoperative endoscopic biopsy: the tumor is located in the upper 1/3 of the stomach (including the esophagogastric junction), and the clinical staging of gastric cancer： Ia and Ib (T1N0M0, T1N1M0, and T2N0M0) (14) according to the eighth edition of the AJCC (15); No distant metastasis was observed on preoperative chest radiograph, abdominal ultrasound, or upper abdominal CT; ASA grade 1-3; Patients without contraindications to surgery; Patients and their families voluntarily signed the informed consent form and participated in the study;

Exclusion Criteria:

Patients diagnosed with primary tumors or distant metastasis; Patients whose tumor is located in the greater curvature side of the stomach; Patients with coagulation dysfunction that could not be corrected; Patients who were diagnosed with viral hepatitis and cirrhosis; Patients who were diagnosed with diabetes mellitus, uncontrolled or controlled with insulin; Patients with organ failure such as heart, lung, liver, brain, and kidney failure; Patients with ascites or cachexia preoperatively in poor general conditions; Patients diagnosed with immunodeficiency, immunosuppression, or autoimmune diseases (such as allogeneic bone marrow transplant, immunosuppressive drugs, SLE, etc.).

Patients refusing to sign the informed consent of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of reflux esophagitis | 12 months after surgery
  The percentage (%) of patients developing postoperative reflux esophagitis after surgery in each group.

SECONDARY OUTCOMES:
incidence of anastomotic leakage | 30 days after surgery
  The percentage (%) of patients developing postoperative anastomotic leakage after surgery in each group.
incidence of anastomotic stenosis | 12 months after surgery
  The percentage (%) of patients developing anastomotic stenosis after surgery in each group.
operative time | 1 day after surgery
  The duration, measured in minutes, spent on reconstructing the digestive tract using different reconstruction methods

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People'S Hospital, Yangzhou, China